CLINICAL TRIAL: NCT01392508
Title: Prospective, Non-interventional, Multi-centre Clinical Study to Assess the Clinical Validity of the Heparin Binding Protein (HBP) Assay for Indicating the Presence, or Outcome, of Severe Sepsis (Including Septic Shock), Over 72 Hours, in Patients With Suspected Infection Following Emergency Department Admission.
Brief Title: IMproved PREdiction of Severe Sepsis in the Emergency Department
Acronym: IMPRESSED
Status: Completed | Type: Observational
Sponsor: Axis Shield Diagnostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-FMHBP-001
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Systemic Inflammatory Response Syndrome (SIRS); Sepsis; Severe Sepsis; Septic Shock
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma (LiHep and citrate)
Oversight: Data Monitoring Committee: No

SUMMARY:
The purposes of this study is to determine whether Heparin Binding Protein (HBP) can be used as a marker of severe sepsis (including septic shock) in patients presenting to the emergency department with suspected infection.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years
* Suspected Infection
* one or more SIRS criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to emergency department with suspected infection
Sampling Method: Probability Sample
Enrollment: 759 (Actual)
Dates: Start 2011-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Linder, Principal Investigator — Skanes Universitetssjukhus I Lund, Sweden; Magnus Paulsson, Principal Investigator — Skanes universitetssjukhuset i Malmo; Patrik Nyberg, Principal Investigator — Universitetssjukhuset i Linkoping; Anna Lange-Jendeberg, Principal Investigator — Universitetssjukhuset i Orebro; Ryan Arnold, Principal Investigator — The Cooper Health System
Locations (5):
- Cooper University Hospital, Camden, New Jersey, United States
- Sweden (4):
  - Universitetssjukhuset i Linkoping, Linköping
  - Skanes Universitetssjukhus i Lund, Lund
  - Skanes Universitetssjukhuset i Malmo, Malmo
  - Universitetssjukhuset i Orebro, Örebro

REFERENCES:
- [Result] Linder A, Arnold R, Boyd JH, Zindovic M, Zindovic I, Lange A, Paulsson M, Nyberg P, Russell JA, Pritchard D, Christensson B, Akesson P. Heparin-Binding Protein Measurement Improves the Prediction of Severe Infection With Organ Dysfunction in the Emergency Department. Crit Care Med. 2015 Nov;43(11):2378-86. doi: 10.1097/CCM.0000000000001265. PMID 26468696